CLINICAL TRIAL: NCT00387803
Title: VENTAK CHF/CONTAK CD Biventricular Pacing Study
Brief Title: Safety and Effectiveness of Cardiac Resynchronization Therapy With Defibrillation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clinicals0010
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2007-01

CONDITIONS: Heart Failure, Congestive; Ventricular Fibrillation; Tachycardia, Ventricular
MeSH Terms: conditions — Heart Failure; Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Cardiac Resynchronization Therapy; Electric Countershock

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy with Defibrillation

SUMMARY:
The purpose of this study was to determine if cardiac resynchronization therapy when combined with defibrillation is safe and effective in the treatment of symptomatic heart failure.

DETAILED DESCRIPTION:
Patients enrolled received a device with cardiac resynchronization therapy (CRT) and defibrillation. Patients were randomized to CRT on or off for up to six months and evaluated for mortality, hospitalization, and functional outcomes including exercise capacity, quality of life, symptomatic status, and echocardiographic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure
* Left ventricular ejection fraction <= 35%
* QRS width >= 120 ms
* Indicated for an implantable cardioverter defibrillator

Exclusion Criteria:

* Indicated for a pacemaker
* Atrial tachyarrhythmias

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 581
Dates: Start 1998-02; Study Completion 2001-08

PRIMARY OUTCOMES:
Composite of all-cause mortality, heart failure hospitalization, and ventricular tachyarrhythmia

SECONDARY OUTCOMES:
Peak VO2
NYHA Class
Six minute walk distance
Quality of life
Echocardiographic measures

CONTACTS AND LOCATIONS:
Overall Officials: Steven Higgins, MD, Principal Investigator — Scripps Memorial Hospital; Leslie A Saxon, MD, Principal Investigator — University of California San Francisco Medical Center; John Boehmer, MD, Principal Investigator — Milton S. Hershey Medical Center; Teresa De Marco, MD, Principal Investigator — University of California San Francisco Medical Center
Locations (1):
- Multiple locations, Saint Paul, Minnesota, United States

REFERENCES:
- [Result] Higgins SL, Hummel JD, Niazi IK, Giudici MC, Worley SJ, Saxon LA, Boehmer JP, Higginbotham MB, De Marco T, Foster E, Yong PG. Cardiac resynchronization therapy for the treatment of heart failure in patients with intraventricular conduction delay and malignant ventricular tachyarrhythmias. J Am Coll Cardiol. 2003 Oct 15;42(8):1454-9. doi: 10.1016/s0735-1097(03)01042-8. PMID 14563591